CLINICAL TRIAL: NCT02321202
Title: Omega-3 Fatty Acid-Based Parenteral Nutrition Improves Postoperative Recovery for Cirrhotic Patients With Liver Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoping Chen, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: bhzhang001
Record Dates: First submitted 2014-12-12; First posted 2014-12-22 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Liver Cancer; Cirrhosis
Keywords: omega-3; Progression; parenteral nutrition
MeSH Terms: conditions — Liver Neoplasms; Fibrosis; Disease Progression; Hyperphagia | interventions — Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): For postoperative parenteral nutrition, only Structolipid applied for 5 consecutive days.
  Interventions: Drug: Structolipid
- Trial group (Experimental): For postoperative parenteral nutrition, Omega-3 Fatty Acid-Based Parenteral Nutrition (20% Structolipid and 10% Omegaven) were applied for 5 consecutive days.
  Interventions: Drug: Omega-3 Fatty Acid-Based Parenteral Nutrition

INTERVENTIONS:
Drug: Omega-3 Fatty Acid-Based Parenteral Nutrition — Glucose, lipid emulsion, amino acids, fat-and water-soluble vitamins as well as electrolytes were compounded in an "All-In-One" manner. 20% Structolipid and 10% Omegaven (ω-3 fatty acid [FA] mainly; Fresenius-Kabi, Germany) were applied to the trial group, but only Structolipid (ω-6 FA mainly) to the control group for 5 consecutive days postoperatively.
  Other Names: trial
  Arms: Trial group
Drug: Structolipid — Glucose, lipid emulsion, amino acids, fat-and water-soluble vitamins as well as electrolytes were compounded in an "All-In-One" manner. 20% Structolipid and 10% Omegaven (ω-3 FA mainly; Fresenius-Kabi, Germany) were applied to the trial group, but only Structolipid (ω-6 FA mainly) to the control group for 5 consecutive days postoperatively.
  Other Names: control
  Arms: Control group

SUMMARY:
The safety and efficacy of ω-3 fatty acid in patients with liver cancer followed hepatectomy is not known. This study provided evidences that ω-3 fatty acid-based parenteral nutrition improved postoperative recovery for cirrhotic patients with liver cancer underwent hepatectomy..

DETAILED DESCRIPTION:
A new lipid emulsion enriched ω-3 fatty acid was manufactured, and was reported avoid hyperinflammatory situations in patients followed major surgery. However, the role of ω-3 fatty acid-based parenteral nutrition for postoperative patients with cirrhosis-related liver cancer is unclear. This study aims to evaluate the safety and efficacy of ω-3 fatty acid-based parenteral nutrition for cirrhotic patients with liver cancer followed hepatectomy.

A prospective randomized controlled clinical trial was conducted for cirrhotic patients with liver cancer underwent hepatectomy between March 2010 and September 2013 in the investigators institution. For postoperative parenteral nutrition, 20% Structolipid and 10% Omegaven were applied to the trial group, while only Structolipid to the control group for 5 consecutive days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* The cirrhotic malnourished patients who were diagnosed as liver cancer preoperatively and underwent hepatectomy were consecutively enrolled.

Exclusion Criteria:

* Contraindication for hepatectomy, including gastrointestinal hemorrhage, severe hemorrhagic disorders, explicit acute nonspecific infectious lesion, overt ascites, Child-Pugh Score C, indocyanine green retention rate at 15min (ICGR15)>30%(12), serum hepatitis B virus (HBV)-DNA>126 copies/ml and serum alanine aminotransferase (ALT) > 2×ULN, serum triglycerides>2.0 mmol/L, circulatory shock, stroke, acute myocardial infarction, renal failure, coma of unknown cause
* Pregnancy
* Age of<18y or>75y
* Performed intraoperative ablation
* Unresectable tumor during operation
* Allergic reactions against fish or egg proteins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
complications (blood test for liver and renal function, urine output, postoperative complications) | 14 days postoperatively
  blood test for liver and renal function, urine output, postoperative complications
hospital stay (time of hospital stay after surgery) | 14 days postoperatively
  the time of hospital stay after surgery

SECONDARY OUTCOMES:
mortality | 30 days postoperatively
  death within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, M.D., Study Chair — Huazhong University of Science and Technology
Locations (1):
- Hepatic Surgery Center of Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Freund HR. Abnormalities of liver function and hepatic damage associated with total parenteral nutrition. Nutrition. 1991 Jan-Feb;7(1):1-5; discussion 5-6. PMID 1802177
- [Background] Carter BA, Shulman RJ. Mechanisms of disease: update on the molecular etiology and fundamentals of parenteral nutrition associated cholestasis. Nat Clin Pract Gastroenterol Hepatol. 2007 May;4(5):277-87. doi: 10.1038/ncpgasthep0796. PMID 17476210
- [Background] Verdery R. Perioperative total parenteral nutrition in surgical patients. N Engl J Med. 1992 Jan 23;326(4):273; author reply 274. No abstract available. PMID 1727984
- [Background] Plauth M, Cabre E, Campillo B, Kondrup J, Marchesini G, Schutz T, Shenkin A, Wendon J; ESPEN. ESPEN Guidelines on Parenteral Nutrition: hepatology. Clin Nutr. 2009 Aug;28(4):436-44. doi: 10.1016/j.clnu.2009.04.019. Epub 2009 Jun 11. PMID 19520466
- [Background] Koller M, Senkal M, Kemen M, Konig W, Zumtobel V, Muhr G. Impact of omega-3 fatty acid enriched TPN on leukotriene synthesis by leukocytes after major surgery. Clin Nutr. 2003 Feb;22(1):59-64. doi: 10.1054/clnu.2002.0592. PMID 12553951
- [Derived] Zhang B, Wei G, Li R, Wang Y, Yu J, Wang R, Xiao H, Wu C, Leng C, Zhang B, Chen XP. n-3 fatty acid-based parenteral nutrition improves postoperative recovery for cirrhotic patients with liver cancer: A randomized controlled clinical trial. Clin Nutr. 2017 Oct;36(5):1239-1244. doi: 10.1016/j.clnu.2016.08.002. Epub 2016 Aug 31. PMID 27614675